CLINICAL TRIAL: NCT05408013
Title: The Prevalence of Insomnia in Patients With Psychiatric Disorders
Status: Recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: Universitätsklinikum Freiburg Klinik für Psychiatrie und Psychotherapie (Unknown); Universitätsklinikum Schleswig-Holstein Klinik für Psychiatrie und Psychotherapie (Unknown); Schlafzentrum Pfalzklinikum Klingenmünster (Unknown); Klinik und Poliklinik für Psychiatrie und Psychotherapie Leipzig (Unknown); Zentralinstitut für Seelische Gesundheit Mannheim (Other); Privatklinik Meiringen (Unknown); Universitätsklinik für Psychiatrie und Psychotherapie, PMU Nürnberg (Unknown); LWL-Klinik Paderborn (Unknown); Klinik für Psychiatrie und Psychotherapie der Universität Regensburg (Unknown); Kompetenzzentrum Schlafmedizin Charité - Campus Benjamin Franklin (Unknown); Klinikum Ingolstadt (withdrawal of participation) (Unknown)
Responsible Party: Principal Investigator, Christoph Nissen, Prof. Dr. med., University of Bern
Other Study IDs: (ID 2020-01992)
Record Dates: First submitted 2021-10-28; First posted 2022-06-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ward patients in psychiatric hospitals: Patients in psychiatric hospitals will be assessed so that the prevalence of insomnia in psychiatric inpatients can be estimated.

SUMMARY:
The primary aim of the proposed project is to investigate the prevalence of insomnia in patients with psychiatric disorders treated as inpatients in psychiatric hospitals in two study sites in Switzerland and nine study sites in Germany. The secondary aim is to investigate whether there are demographic or disorder specific parameters that influence the prevalence of insomnia in patients with psychiatric disorders.

DETAILED DESCRIPTION:
QUALITY ASSURANCE PLAN & SOURCE DATA VERIFICATION

For quality assurance the Ethics Committee may visit the research sites. For each study participant, a paper based case report form (CRF) will be maintained. CRFs will be kept current to reflect subject status at each phase during the course of study. Data for statistical analysis will be stored in an electronic database. Data will be transferred manually from the paper CRF to the electronic data base. As for the paper based CRF, the data stored electronically will not contain any personal information by which the participant can be identified. Only trained project personnel will be authorized for entries into the electronic database and authorized persons will be identifiable for every entry they made. Routinely collected data during daily clinical practice will be transferred to the participant CRF (e.g. diagnoses and medication).

DATA DICTIONARY

BASEC, Business Administration System for Ethical Committees CRF, Case report form FOPH, Federal Office of Public Health HRA, Human Research Act HRO, Ordinance on Human

STANDARD OPERATING PROCEDURE The recruitment of the study participants is consecutive. In all study sites, all newly admitted patients will be registered on a list each day. This list will be available for the study physicians. From this list, patients who are visibly not eligible (involuntary stay, under custody) will be deleted. Depending on the capacities of the study physicians, within three days after admission, 1-15 patients will be selected from the patients remaining on the list per day. The selected patients will be asked whether they agree to participate in the study.

The overall project duration will be 12 months starting the 1st of July 2021 until the end of June 2022. The patients will be screened according to the inclusion and exclusion criteria. The study investigator will then hold one session of 20 to 60 minutes with each participant filling out the following questionnaires:

* The study information and the informed consent
* The informed consent about the further use of the patient data
* Demographic data and general patient documentations
* PSQI: Pittsburgh sleep quality index
* ISI: Insomnia severity index
* The Epworth Sleepiness Scale
* SF-12: Short form 12 questionnaire about the subjective health status
* PHQ-9: Patient health questionnaire 9
* Fatigue Severity Screening

Participants will be withdrawn from the study immediately if there are any concerns about the participants' safety. Participants can also choose to withdraw from the study at any time, and are not required to provide their reason for withdrawing from the study. Coded data acquired before withdrawal will be analyzed as described in the participant information sheet.

If a serious event occurs, the research project will be interrupted and the Ethics Committee notified on the circumstances via BASEC within 7 days according to HRO Art. 21 .

SAMPLE SIZE ASSESSMENT & STATISTICAL ANALYSIS PLAN

In Table 1 in the study protocol which is attached in the documents section, the 95%- confidence intervals for prevalence in the range from 15% (p=0.15) to 25% (p=0.25) can be seen for sample sizes of n= 200, n= 250, n=300 and n= 500 patients. In consideration of the accuracy of the estimation of varying prevalence, the planned study aims to investigate 500 psychiatric inpatients. The named sample size will be sufficient to estimate prevalence rates with sufficient power.

PLAN FOR MISSING DATA Dropouts will be replaced by recruitment of new participants until the target sample size has been achieved.

ELIGIBILITY:
Inclusion Criteria:

* patients who suffer from a psychiatric disorder according to the DSM-5 and who are currently treated as inpatients in one of these psychiatric hospitals:

  2 swiss study sites: Universitäre Psychiatrische Dienste in Bern, Privatklinik Meiringen.

  9 german study sites: Freiburg, Ingolsatdt, Kiel, Klingenmünster, Leipzig, Mannheim, Nürnberg, Paderborn, Regensburg

Exclusion Criteria:

* Age under 18 years
* involuntary stay at the clinic
* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffer from a psychiatric disorder according to the DSM-5 and who are currently treated as inpatients in a psychiatric hospital
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Disorder | Day 1
  The prevalence of insomnia disorder will be assessed at a one-time point per patient during a study session with a clinician.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Nissen, Prof. Dr. med, Principal Investigator — Sleep Research in Psychiatry
Locations (1):
- Universitäre Psychiatrische Dienste Bern (Upd), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Participant data that underlie the results reported in the future article after deidentification will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: In the end of the study the coded data will be sent to Berlin and used for result calculations
Access Criteria: Encrypted data will be sent via secure mails to heidi.danker-hopfe@charite.de. The code to open the encrypted data will be sent via a separate mail. The methods are conform with the regulations of the ethics commission of Switzerland and Germany.

REFERENCES:
- [Background] Seow LSE, Verma SK, Mok YM, Kumar S, Chang S, Satghare P, Hombali A, Vaingankar J, Chong SA, Subramaniam M. Evaluating DSM-5 Insomnia Disorder and the Treatment of Sleep Problems in a Psychiatric Population. J Clin Sleep Med. 2018 Feb 15;14(2):237-244. doi: 10.5664/jcsm.6942. PMID 29394962

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT05408013/Prot_SAP_000.pdf